CLINICAL TRIAL: NCT04970966
Title: Efficacy of PuraSinus Versus Bioresorbable Nasal Dressings in Improving Patient Comfort During Postoperative Debridements
Brief Title: Efficacy of PuraSinus Versus Bioresorbable Nasal Dressings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Kevin Hur, Principal Investigator, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-03390
Record Dates: First submitted 2021-07-11; First posted 2021-07-21 (Actual); Results first posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Sinus Disease; Surgery
Keywords: sinus surgery; chronic rhino sinusitis

STUDY DESIGN:
Intervention Model Description: Intra-patient control
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PuraSinus (Experimental): Placement of PuraSinus in ethmoid cavity following ESS
  Interventions: Device: PuraSinus
- Bioresorbable Nasal Dressing (Active Comparator): Placement of bioresorbable nasal dressing (PosiSep X) in ethmoid cavity following ESS
  Interventions: Device: Bioresorbable Nasal Dressing

INTERVENTIONS:
Device: PuraSinus — A randomized ethmoid cavity in the patient will have PuraSinus applied to the ethmoid cavity after completion of an endoscopic total ethmoidectomy.
  Arms: PuraSinus
Device: Bioresorbable Nasal Dressing — PosiSep X will be applied to the ethmoid cavity after completion of an endoscopic total ethmoidectomy.
  Arms: Bioresorbable Nasal Dressing

SUMMARY:
Postoperative care of patients undergoing endoscopic sinus surgery (ESS) is important both to minimize discomfort for the patients and to obtain the optimal long-term outcomes. Postoperative sinonasal cavity debridement has been advocated to prevent potential synechiae and sinus ostial stenosis, as well as to improve patient symptoms. Removal of old blood, nasal secretions, crusting, and unabsorbed packing are thought to reduce the inflammatory load, minimize potential for scarring, and allow for improved access of topical medications. However, the debridement procedure can cause bleeding, pain, and discomfort which may interfere with the effective execution of postoperative care.

PuraSinus is a novel topical haemostatic agent based on nanotechnologies in the form of a transparent hydrogel suitable for endoscopic use and for which the use in sinonasal surgery could achieve these various goals. The potential of PuraSinus to enhance endoscopic mucosal wound healing may play a role in optimizing patient comfort during postoperative debridements after ESS. However, clinical evidence on its effectiveness in ESS is limited.

The investigators aim to perform a randomized controlled trial to evaluate the efficacy of PuraSinus in improving patient comfort during postoperative debridements among patients who underwent ESS.

DETAILED DESCRIPTION:
Postoperative formation of adhesions, scarring, synechiae, ostial stenosis and edema are major concerns often addressed by the placement of bioresorbable packing intraoperatively. Bioresorbable packing has been demonstrated to decrease the incidence of adhesions and bleeding while improving patient comfort compared to no packing at all. However, bioresorbable nasal dressings oftentimes have not dissolved by the time of the first postoperative debridement 1-2 weeks after the surgery and therefore need to be removed. The removal of bioresorbable packing during postoperative debridements is usually an uncomfortable experience for the patient. An ideal nasal dressing would optimize both patient comfort as well as wound healing.

This is a prospective randomized controlled multicenter study at the University of Southern California and Northwestern University that will enroll at least 30 participants who satisfy criteria to compare the efficacy of PuraSinus versus standard of care in patients undergoing endoscopic sinus surgery. The study will utilize an intra-patient control design to assess the safety and efficacy of PuraSinus compared to bioresorbable packing on the contralateral side. The study patients will undergo PuraSinus placement in one nasal cavity following traditional endoscopic sinus surgery. The study is blinded, meaning that patients will be blinded throughout the study duration to which side received PuraSinus placement. The independent surgeon performing review of the video-endoscopies will also be blinded to which side received PuraSinus.

The patient will undergo follow-up assessments including endoscopic examination at three (3) post-operative visits at week 1, week 4, and week 12. A postoperative endoscopic debridement of the ethmoid cavities will be performed bilaterally at week 1. Primary and secondary outcomes will be assessed during the postoperative visits.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient has a clinical indication for and has consented for primary or revision bilateral ESS and had evidence of ethmoid disease bilaterally (Lund-Mackay score at least 1 on each side).
* Diagnosed with CRS based on American Academy of Otolaryngology - Head and Neck Surgery guidelines

Exclusion Criteria:

* Patient has a known history of immune deficiency such as immunoglobulin G or A subclass deficiency, or Human Immunodeficiency Virus (HIV).
* Patient has concurrent condition requiring active chemotherapy and/or immunotherapy management for the disease (e.g. cancer, HIV, etc.)
* Patient has clinical evidence of disease or condition expected to compromise survival or ability to complete follow-up assessments during the 90 day followup period.
* Patient is currently participating in another clinical trial.
* Patient has a known coagulation disorder.
* Patient is allergic to shellfish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-05-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Keck Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a split-person (within-participant) design: each participant contributed one ethmoid cavity to the Hydrogel arm and the contralateral cavity to the Chitosan arm. Therefore, the same participants are counted in both arms within a Milestone row, which is expected.
Units Other Than Participants: Right or Left Ethmoid Cavity
Groups:
- Hydrogel (Treatment Side): Participant had hydrogel placed in ethmoid cavity.
- Chitosan-based Polymer (Control): Participant had chitosan-based polymer placed in ethmoid cavity
Period: Week 1 Follow-up
Arm/Group | Hydrogel (Treatment Side) | Chitosan-based Polymer (Control)
Started | 30; 30 Right or Left Ethmoid Cavity | 30; 30 Right or Left Ethmoid Cavity
Completed | 30; 30 Right or Left Ethmoid Cavity | 30; 30 Right or Left Ethmoid Cavity
Not Completed | 0; 0 Right or Left Ethmoid Cavity | 0; 0 Right or Left Ethmoid Cavity
Period: Week 4 Follow-up
Arm/Group | Hydrogel (Treatment Side) | Chitosan-based Polymer (Control)
Started | 30; 30 Right or Left Ethmoid Cavity | 30; 30 Right or Left Ethmoid Cavity
Completed | 30; 30 Right or Left Ethmoid Cavity | 30; 30 Right or Left Ethmoid Cavity
Not Completed | 0; 0 Right or Left Ethmoid Cavity | 0; 0 Right or Left Ethmoid Cavity
Period: Weed 12 Follow-up
Arm/Group | Hydrogel (Treatment Side) | Chitosan-based Polymer (Control)
Started | 30; 30 Right or Left Ethmoid Cavity | 30; 30 Right or Left Ethmoid Cavity
Completed | 28; 28 Right or Left Ethmoid Cavity | 28; 28 Right or Left Ethmoid Cavity
Not Completed | 2; 2 Right or Left Ethmoid Cavity | 2; 2 Right or Left Ethmoid Cavity

BASELINE CHARACTERISTICS:
Population: All randomized participants who underwent bilateral total ethmoidectomy.
Groups:
- Participants: All randomized participants who underwent bilateral total ethmoidectomy
Arm/Group | Participants
Number analyzed (Participants) | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48.5 [38 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
History of Endoscopic Sinus Surgery [Count of Participants; unit: Participants] | 6
Nasal Polyps [Count of Participants; unit: Participants] | 11
Allergic Rhinitis [Count of Participants; unit: Participants] | 10
Asthma [Count of Participants; unit: Participants] | 6
Diabetes [Count of Participants; unit: Participants] | 4

OUTCOME MEASURES:

1. Primary Outcome: Pain During Debridement
Description: Patient-reported pain visual analogue scale during postoperative debridement of ethmoid cavity. The minimum score is 1, which reflects no pain, and the maximum score is 10, which reflects an extreme amount of pain.
Time Frame: 1 week after surgery
Measure: Median (Inter-Quartile Range); unit: Pain Score
Arm/Group | Hydrogel (Treatment Side) | Chitosan-based Polymer (Control)
Number analyzed (Participants) | 30 | 30
Pain Score | 4 [2.5 to 5.5] | 5 [4 to 6]

2. Secondary Outcome: Debridement Time
Description: Time required to perform sinonasal cavity debridement for ethmoid cavity 1 week after surgery
Time Frame: 1 week after surgery
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Hydrogel (Treatment Side) | Chitosan-based Polymer (Control)
Number analyzed (Participants) | 30 | 30
minutes | 1.96 [1.05 to 2.89] | 1.57 [1.08 to 2.06]

3. Secondary Outcome: Number of Participants With Mucosal Edema
Description: Mucosal edema was assessed via endoscopic examination at 4 weeks postoperatively. Edema was recorded as present or absent based on investigator visual assessment using standard postoperative sinus endoscopy criteria
Time Frame: 4 weeks after surgery
Population: Data were available for 28 participants per arm at this time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrogel (Treatment Side) | Chitosan-based Polymer (Control)
Number analyzed (Participants) | 28 | 28
Participants | 24 | 24

4. Secondary Outcome: Number of Participants With Postoperative Adhesions at 12 Weeks
Description: Adhesions were assessed during endoscopic examination at 12 weeks postoperatively. Presence of adhesions was determined by direct visualization of scar bands between the middle turbinate and lateral nasal wall.
Time Frame: 12 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrogel (Treatment Side) | Chitosan-based Polymer (Control)
Number analyzed (Participants) | 28 | 28
Participants | 1 | 1

5. Secondary Outcome: Number of Participants With Postoperative Bleeding at Week 1 Debridement
Description: Bleeding was evaluated during the week 1 postoperative debridement visit. Presence of bleeding was recorded if any mucosal bleeding was visualized on nasal endoscopy in the ethmoid cavity.
Time Frame: 1 week after surgery
Population: Two participants did not have evaluable endoscopic data at this time point and were excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrogel (Treatment Side) | Chitosan-based Polymer (Control)
Number analyzed (Participants) | 28 | 28
Participants | 23 | 23

6. Secondary Outcome: Number of Participants With Greater Than 50% Residual Dressing in Ethmoid Cavity at Week 1
Description: Residual bioresorbable dressing material in the ethmoid cavity was assessed endoscopically at 1 week. Greater than 50% residual material was recorded when more than half of the originally placed dressing remained visible.
Time Frame: 1 week after surgery
Population: Two participants did not have evaluable endoscopic data at this time point and were excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrogel (Treatment Side) | Chitosan-based Polymer (Control)
Number analyzed (Participants) | 28 | 28
Participants | 9 | 13

7. Secondary Outcome: Number of Participants Requiring Additional Postoperative Intervention by Week 4
Description: The need for further intervention postoperatively 4 weeks after surgery as evaluated by an independent blinded reviewer of the video-endoscopy
Time Frame: 4 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrogel (Treatment Side) | Chitosan-based Polymer (Control)
Number analyzed (Participants) | 30 | 30
Participants | 1 | 4

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, up to 12 weeks
Groups:
- Hydrogel (Treatment Side): Participants who received hydrogel in at least one ethmoid cavity
- Chitosan-based Polymer (Control): Participants who received chitosan dressing in at least one ethmoid cavity
Arm/Group | Hydrogel (Treatment Side) | Chitosan-based Polymer (Control)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT04970966/Prot_SAP_000.pdf